CLINICAL TRIAL: NCT01507675
Title: Burden, Belonging, and Response to Pain in Veterans
Status: Withdrawn | Type: Observational
Why Stopped: Study should not have been listed on ClinicalTrials
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: COMIRB 11-0948
Record Dates: First submitted 2011-12-09; First posted 2012-01-11 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Suicide
Keywords: suicide; psychometric properties; military; veterans; Interpersonal needs questionnaire; Acquired capability for suicide; mental health; Survey of Life Principles; Risk assessment
MeSH Terms: conditions — Suicide; Psychological Well-Being

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Military Veterans: Participants will be recruited from the Denver VA Medical Center (DVAMC), regardless of clinic.

SUMMARY:
The primary purpose of the current study is to rigorously test the psychometric properties of the INQ-12 and ACSS (Van Orden et al., 2008) in Veterans, something which has not been done to date. Factor structure, internal consistency, convergent and discriminant validity will all be assessed. Secondary goals are to determine if burdensomeness, failed belongingness, and acquired capability are distinct versus overlapping constructs and whether or not values mediate the relationship between reasons for living and suicide risk. Lastly, the inclusion of the Beck Scale for Suicidal Ideation (BSS) allows us to analyze participants' responses to explore whether or not participants can be grouped into those who want to die by suicide because they want to escape their problems and those who want to die to influence other people.

DETAILED DESCRIPTION:
Suicide is a significant problem among Veterans of the U.S. Military. Katz (2007) reported that there were 144 suicides among Veterans who served in Operation Enduring Freedom (OEF) and/or Operation Iraqi Freedom (OIF) from 2002-2005. There is no nationwide surveillance system that tracks Veteran suicides. However, the National Violent Death Reporting System (NVDRS) created in 2003 by the Centers for Disease Control and Prevention (CDC) with the purpose of gathering thorough information about suicides and other violent deaths allows researchers to reasonably extrapolate national suicide rates for Veterans. A CDC report (2006) based on NVDRS data estimated that approximately 6,500 veterans from all wars die by suicide each year, accounting for approximately 20% of suicides per year nationwide. While much is known about risk factors for suicide (e.g., Beck, Steer, Kovacs, & Garrison, 1985; Jobes & Mann, 1999) such information has little clinical utility for predicting whether or not an individual is likely to die by suicide in the near-term. One of the few attempts to address this issue is the interpersonal-psychological theory of suicide (Joiner, 2005). The interpersonal psychological theory proposes that people die by suicide for three reasons: (1) they perceive themselves as a burden to others; (2) they experience a profound feeling of disconnectedness from others, what Joiner (2005) calls ''thwarted belongingness'' (p. 118); and (3) they have become habituated to the fear and physical pain inherent in a suicidal act by repeatedly enduring painful and provocative situations, whether through such experiences as repeated suicide attempts, other physically painful experiences, or frequent exposure to danger. Importantly, all three factors must be present for a suicide to occur, according to the interpersonal-psychological theory; together, these three characteristics are ''proximal, causal, interactive risk factors'' (Van Orden, Witte, Gordon et al., 2008a, p. 72). Components of the theory have been tested in adults (Joiner, Pettit, Walker, Voelz, Cruz, & Rudd, 2002; Joiner & Rudd, 2000), college students, and adolescents (Joiner, Rudd, Rouleau, & Wagner, 2000). However, research has only begun to explore whether the theory applies to Veterans (Cornette, Deboard, Clark, Holloway, Brenner, Gutierrez, et al., 2007; Cornette, deRoon-Cassini, Joiner, & Proescher, 2006). Brenner et al. (2008) conducted a qualitative study of OEF/OIF Veterans which found relevance of the theory to their experiences. In particular, themes emerged around combat as a context for exposure to painful stimuli, perceptions of burdensomeness, and failed belongingness. This theory shows promise for designing prevention and clinical intervention strategies for Veterans, but more data are needed on which to base such work. To facilitate testing the interpersonal-psychological theory of suicide, Joiner and colleagues have developed several instruments (Bender, Gordon, & Joiner, 2007; Bryan, Morrow, Anestis, & Joiner, 2010; Van Orden,Witte, Gordon et al., 2008a). The Interpersonal Needs Questionnaire (INQ) taps into the constructs of thwarted belongingness and perceived burdensomeness. The Acquired Capability for Suicide Scale (ACSS; Van Orden et al., 2008) measures fearlessness about suicide. The current study will focus on the 12-item version of the INQ (INQ-12; Van Orden, Witte, Gordon, Bender, & Joiner, 2008a) recently validated by Freedenthal, Lamis, Osman, Kahlo, and Gutierrez (2011). This measure contains seven items that assess perceived burdensomeness and five items that assess belongingness. An example of a burdensomeness item in the INQ-12 is, ''These days, I think I have failed the people in my life''. An example of a belongingness item is, ''These days, other people care about me''. The ACSS is a 20-item measure rated on a scale of 1 (not at all like me) to 5 (very much like me). Sample items include, "I am not at all afraid to die" and "I can tolerate a lot more pain than most people". Van Orden et al. report acceptable convergent and discriminant validity. The authors also reported a strong negative correlation with the fear of suicide subscale on the Reasons for Living Inventory (RFL; Linehan, Nielsen, & Chiles, 1983) and a positive correlation with the courage to kill oneself item on the Beck Scale for Suicide Ideation (BSS; Beck & Steer, 1991). Bender, Gordon, Bresin, and Joiner (2011) reported acceptable internal consistency as well. However, formal psychometric studies of the ACSS have yet to be conducted. Joiner (2005) describes burdensomeness, failed belongingness and acquired capability as separate constructs, with the INQ-12 and ACSS designed to assess each independently. However, for purposes of explaining whether a given individual is likely to die by suicide, Joiner et al. (2009) explain that the first two constructs together create the desire for death and that the third is necessary for a person to engage in potentially lethal self-harm behavior. Therefore, a complex interaction between the three is proposed. Support for this interaction was found by Joiner et al. in two independent samples, one community sample of young adults and a second drawing on archival data from active duty military personnel being treated for a recent significant suicide-related event (e.g., serious ideation or attempt). A major limitation of this study was that measures of the constructs differed, making it somewhat difficult to determine what was being assessed in the two samples. Additionally, in their psychometric examination of the INQ-12 Freedenthal and colleagues (2011) found evidence of an overarching factor uniting the two subscales of burdensomeness and failed belongingness. Assessing for suicide risk is a key element of the clinical management of high-risk individuals (Gutierrez et al., 2009), but is only the first step. To adequately select appropriate interventions clinicians must know what is driving an individual's suicidality (Jobes, 2006) and also what factors are keeping the person from acting on their thoughts and urges. This information better helps the clinician and client to develop strategies aimed at creating (or rediscovering) what makes life worth living; focusing on plans, goals, and hope for the future (Jobes, Comtois, Brenner, & Gutierrez, 2011). Historically, the RFL (Linehan et al., 1983) has been one of the primary measures of protective factors against suicide, and indeed has shown great utility. A potentially related area of study is the role of one's values. The consciously chosen way in which an individual lives her life, the driving force behind her actions, and the desired outcomes of her behaviors define what an individual values (Luoma, Hayes, & Walser, 2007). Helping clients live lives consistent with their values provides purpose and meaning, gives direction to their choices, and allows them to set reasonable, flexible goals likely to motivate meaningful action (Luoma et al.). Accomplishing these things should greatly facilitate reducing an individual's risk of suicide, since it answers the fundamental existential question "why is life worth living?" Ciarrochi and Bailey (2008) created the Survey of Life Principles to assess values, and provide preliminary support for its use in their manual.

ELIGIBILITY:
Inclusion Criteria:

* Military veteran
* 18 or older
* Ability to respond to questions regarding the informed consent

Exclusion Criteria:

* Active-duty military
* Non-English speaking
* Inability to respond to questions regarding the informed consent procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from all individuals eligible to receive care at the Denver VA Medical Center (DVAMC), regardless of clinic.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Internal consistency reliability. | two years
  The internal consistency reliability statistics will be calculated for all study variables to confirm the measures are reliable.
Convergent validity. | two years
  Convergent validity of the Interpersonal Needs Questionnaire (INQ) will be determined by examining the correlation between it and the other study measures.
Convergent validity. | two years
  Convergent validity of the acquired capability of suicide scale (ACSS) will be determined by correlating it with all other measures.

SECONDARY OUTCOMES:
Discriminant validity. | two years
  Discriminant validity of the interpersonal needs questionnaire (INQ) will be determined by examining correlations with measures of unrelated constructs.
Suicide risk. | two years
  Examine the effects of scores on the SLP on the relationship between reasons that people have for living and the potential for engaging in at-risk behavior.
Discriminant validity | two years
  Examine the discriminant validity of the acquired capability for suicide scale (ACSS) by examining correlations between it and measures of unrelated constructs.

CONTACTS AND LOCATIONS:
Overall Officials: Peter M. Gutierrez, PhD, Principal Investigator — Clinical Research Psychologist VA VISN 19 MIRECC
Locations (1):
- Va Visn 19 Mirecc, Denver, Colorado, United States

REFERENCES:
- See also: The mission of the VISN 19 MIRECC is to study suicide with the goal of reducing suicidality in the veteran population. — http://www.mirecc.va.gov/visn19